CLINICAL TRIAL: NCT01953315
Title: A Phase 1 Pilot Safety and Feasibility Study of Muscle Progenitor Cell (MPC) Therapy for Urinary Incontinence
Brief Title: Muscle Progenitor Cell Therapy for Urinary Incontinence
Acronym: MPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00023616
Record Dates: First submitted 2013-08-27; First posted 2013-09-30 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2018-01

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, muscle progenitor cells, MPCs
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Muscle Progenitor Cells (Experimental): Autologous MPCs, administered via a single, direct injection into the bladder neck sphincter region
  Interventions: Biological: Autologous Muscle Progenitor Cells

INTERVENTIONS:
Biological: Autologous Muscle Progenitor Cells — Autologous MPCs, administered via a single, direct injection into the bladder neck sphincter region
  Other Names: MPCs

SUMMARY:
This study is designed to evaluate the safety of muscle progenitor cells (MPCs) for the treatment of urinary incontinence due to incompetent outlet (bladder neck/urethra).

DETAILED DESCRIPTION:
Eligible subjects with a diagnosis of urinary incontinence who give consent to take part will undergo a biopsy of the muscle from the inner thigh under anesthesia. The muscle sample will be cultured and expanded for approximately 6 weeks. The product, composed of autologous, ex vivo-expanded muscle progenitor cells (MPCs) in suspension, will be delivered via targeted injection into the bladder neck sphincter region using either an endoscopic needle via a cystoscope or periurethral injection under ultrasound guidance. All subjects will be followed at 1 week, 6 weeks, 3 months, 6 months and 12 months post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients who are not pregnant or lactating/breast-feeding and must be either not sexually active, surgically sterilized, or must be practicing an effective method of birth control as determined by the investigator (e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy)
* Patients between the ages of 18 and 75 years
* Patients with positive diagnosis of urinary incontinence due to sphincter insufficiency caused by acquired (e.g., stress urinary incontinence) and/or congenital (bilateral ectopic ureters with incompetent bladder neck; or female epispadias with or without bladder exstrophy) conditions.
* Patients with cystometric capacity of bladder > 100 ml
* Patients with normal renal function
* Patients with a history of primary incontinence

Exclusion Criteria:

* Patients with a history of hypercontractile bladder, non-compliant bladder, hydronephrosis or neurogenic bladder
* Patients with an active urinary tract infection as evidenced by positive urine culture
* Patients who are taking medication that affect urination (e.g. medically necessary, stable drugs) such as prescription drugs, over-the-counter drugs, or dietary supplements, including herbal supplements and those taken with teas
* Patients requiring concomitant use of or treatment with immunosuppressive agents
* Patients with a history of systemic conditions, including but not limited to HIV, diabetes and chronic liver disease (including Hepatitis B or C), that the Investigator believes may jeopardize the safety of the patient to participate in the study
* Patients with evidence or diagnosis of any primary muscle disease or coagulation disorder (including concomitant anti-coagulation therapy at enrollment)
* Patients who have been treated with any other investigational drug or participated in any investigational study within 30 days prior to enrollment in this study
* Patients with urinary incontinence other than the categories being investigated
* Patients with significant (>grade 2) pelvic organ prolapse (e.g., cystocele, rectocele)
* Patients with vaginal prolapse beyond introitus
* Patients with neurological disorders (e.g., multiple sclerosis, Parkinson's disease)
* Patients with abnormal bladder capacity (i.e., less than 100 cc)
* Patients with abnormal urologic conditions, including post-void residual, urethral stricture and bladder neck contracture, spastic bladder, vesicoureteral reflux, bladder stones, bladder tumors, hydronephrosis, other renal impairment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related serious adverse events and the incidence of protocol defined treatment or procedure related adverse events | 12 months
  the subject/biopsy/treatment site will be monitored for signs of bleeding, infection, continued pain, prolonged hospitalization

SECONDARY OUTCOMES:
change in Incontinence Assessment by pad test | baseline, 3, 6, and 12 months post-injection
  Subjects will undergo 1 hour and 24 hour pad tests (pads are weighed)at baseline which are compared to the tests post-injection treatment
change in Number of incontinence episodes and pads used per day | baseline, 3, 6 and 12 months post-injection treatment
  through Voiding diaries, the number of incontinence episodes and pads used per day are compared to baseline
change in Urogenital distress and quality of life | baseline, 3, 6 and 12 months post-injection treatment
  subjects will complete the Urinary Incontinence and Quality of Life questionnaires and the baseline results will be compared to the 3, 6 and 12 months post injection results.

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Badlani, MD, Principal Investigator — Wake Forest School of Medicine, Dept. of Urology
Locations (2):
- United States (2):
  - Wake Forest Urology Clinic, Winston-Salem, North Carolina
  - Wake Forest Institute for Regenerative Medicine (WFIRM), Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No